CLINICAL TRIAL: NCT04541160
Title: Ultra-low Dose Chest Computed Tomography: a Rule-out Tool for Community-acquired Pneumonia
Status: Completed | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Other Study IDs: 3083
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2017-10

CONDITIONS: Pneumonia; Diagnoses Disease
Keywords: pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Suspected community-acquired pneumonia patients: Suspected community-acquired pneumonia patients that will be evaluated by an imaging method
  Interventions: Diagnostic Test: CR; Diagnostic Test: ULDCT

INTERVENTIONS:
Diagnostic Test: CR — Lung imaging evaluation performed with CR
Diagnostic Test: ULDCT — Lung imaging evaluation performed with ULDCT

SUMMARY:
This is a randomized study that sought to compare the rule-out capacity and antibiotics prescriptions associated with two different diagnostic imaging strategies (ultra-low-dose chest computed tomography versus chest radiography) in a group of healthy adults presenting to the emergency department (ED) with suspected community-acquired pneumonia (CAP).

DETAILED DESCRIPTION:
Between October 2017 and December 2018, we prospectively enrolled consecutive adult patients with suspected community-acquired pneumonia based on at least one respiratory symptom and focal auscultatory findings and at least one sign related to infection, for whom no definitive diagnosis was possible by clinical judgment.

Eligible patients were randomly assigned to their imaging evaluation in a 1:1 ratio to either ultra-low-dose chest computed tomography (ULDCT) or the standard evaluation strategy using conventional chest radiography (CR).

This study sought to compare the rule-out capacity and antibiotics prescriptions associated with those two different diagnostic imaging strategies (ULDCT versus CR) in a group of healthy adult patients presenting to the ED with suspected CAP.

ELIGIBILITY:
Inclusion Criteria:

* Suspected CAP;
* At least one respiratory symptom (new or increasing cough, expectoration, dyspnea or chest pain) and
* At least one symptom related to infection (fever ≥ 38°C, chills, sweating, myalgia, mental confusion or headache) and
* Focal auscultatory findings during physical examinations (crackling rales)
* No definitive diagnosis possible by clinical judgment.

Exclusion Criteria:

* Score in at least one clinical part of the CURB-65 or PSA scores
* Clinical diagnosis of rhinosinusitis and acute nasopharyngitis and who had already been treated with antimicrobial therapy for this episode of disease
* pregnancy;
* the presence of other respiratory diseases such as chronic obstructive pulmonary disease (COPD), asthma, interstitial lung disease, chronic diseases or other chronic airway conditions;
* diagnosis of congestive heart failure;
* body mass index (BMI) greater than 30;
* inability to hold the breath for at least 10 seconds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 211 patients were included from the 237 eligible ones. Sixteen patients refused to sign the informed consent form and five were excluded due to technical errors during image acquisition. Two patients exhibited BMIs higher than 35 and did not fulfil the inclusion criteria; three patients could not be reached for follow-up.
  Among the 211 patients included, 98 (46.45%) were imaged by CR and 113 (53.55%) by ULDCT. There were no significant differences among patients in the CR and ULDCT groups concerning age, gender, height, weight, and BMI.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Community-acquired pneumonia rule-out capability | 1 month
  Number of Participants for whom ULDCT could diagnose absence of imaging signs of pneumonia
Antibiotics prescription | immediate
  Number of Participants for whom antibiotics were prescribed to treat bacterial pneumonia

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data (IPD) available to other researchers.